CLINICAL TRIAL: NCT03502681
Title: Phase 1b Clinical Trial of Eribulin Mesylate and the PD-L1 Monoclonal Antibody, Avelumab, in Cisplatin Ineligible Metastatic Urothelial Cell Cancer Patients
Brief Title: A Study Combining Eribulin Mesylate With Avelumab in Cisplatin Ineligible Metastatic Urothelial Cell Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funder Decision
Sponsor: Monika Joshi, MD (Other)
Collaborators: Pfizer (Industry); Eisai Inc. (Industry); Big Ten Cancer Research Consortium (Other)
Responsible Party: Sponsor-Investigator, Monika Joshi, MD, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-GU16-051
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Results first posted 2020-07-09 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Urothelial Cell Cancer
Keywords: Cisplatin-Ineligible; Avelumab; PD-L1 Monoclonal Antibody; Eribulin Mesylate
MeSH Terms: interventions — eribulin; avelumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Maximum tolerated dose (MTD) cohort (Experimental): The initial 9-12 patients (MTD cohort) will be enrolled to determine safety of avelumab in combination with eribulin mesylate.
  Upon determination of maximum tolerated dose (MTD), 12 additional patients will be enrolled in an expansion cohort (efficacy cohort) to determine objective response rate (ORR) at 6 months.
  Interventions: Drug: Eribulin Mesylate; Drug: Avelumab

INTERVENTIONS:
Drug: Eribulin Mesylate — Days 1, 15
  Eribulin mesylate:
  Dose level -1: 0.7mg/m^2;
  Dose level 0: 1.1 mg/m^2;
  Dose level +1: 1.4 mg/m^2
  Other Names: Halaven
Drug: Avelumab — Days 1, 15 Avelumab (10mg/kg)
  Other Names: MSB0010718C; BAVENCIO

SUMMARY:
This is a single arm, open-label phase Ib study of combining eribulin mesylate with avelumab. The initial 9-12 patients (MTD cohort) will be enrolled to determine safety of avelumab in combination with eribulin mesylate. Upon determination of maximum tolerated dose (MTD), 12 additional patients will be enrolled in an expansion cohort (efficacy cohort) to determine ORR at 6 months.

DETAILED DESCRIPTION:
Dose Escalation Plan:

A standard "3+3" design will be used to determine the MTD of eribulin with avelumab.

The maximum tolerated dose is the dose of eribulin combined with avelumab with dose limiting toxicity of 0-1 of 6 patients in the first cycle of combination therapy. After the MTD has been determined, an additional 12 patients will be enrolled in an expansion cohort at the MTD to evaluate the efficacy of this combination.

After determination of MTD for eribulin mesylate, an additional 12 patients will be enrolled on the expansion cohort. Subjects on the expansion cohort will be assessed for adverse events but will not be assessed for DLTs.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0-2 at the time of enrollment.
* Life expectancy of >12 weeks.
* Stage IV patients either locally advanced node positive (these patients must have N3 disease) or metastatic-M1 positive urothelial cancer of bladder and upper tract.
* Histologically proven urothelial carcinoma of bladder with predominant transitional cell component. Adenocarcinoma, squamous cell differentiation, or other atypical histology (such as plasmacytoid or sarcomotoid) of the bladder will be allowed on the study, provided they form <50% of the histology.
* Presence of measurable disease per RECIST v1.1 for solid tumors.
* Patients who are cisplatin ineligible defined by the presence of one or more of the following:

  * Impaired renal function (GFR ≥ 30 but ≤ 60 cc/min). GFR should be assessed by direct measurement (i.e. creatinine clearance or ethylenediaminetetra-acetate) or, if not available, by calculation from serum/plasma creatinine by Cockroft-Gault equation.
  * Grade ≥ 2 Hearing Loss (hearing loss measured by audiometry of 25 dB at two contiguous frequencies)
  * Grade ≥ 2 peripheral neuropathy (Please note that for enrollment on this trial patients must have peripheral neuropathy grade 2 or lower)
  * ECOG Performance Status of 2
  * NYHA Class III-IV CHF (Please note that for enrollment on this trial patients must have Ejection Fraction of >35% measured on ECHO)
* Patients must be treatment naïve for metastatic disease. Use of chemotherapy in neoadjuvant or adjuvant form is allowed provided the time period between last dose of treatment and enrollment is >12 months and subjects must have recovered from all reversible toxic effects of the regimen (other than alopecia) to ≤Grade 1 or baseline.
* Demonstrate adequate organ function as defined below; all screening labs to be obtained within 28 days prior to study registration:

Hematological:

* Platelet ≥ 100K/mm^3
* Absolute Neutrophil Count (ANC) ≥ 1.5 K/mm^3
* Hemoglobin (Hgb) ≥ 9 g/dL

Renal:

* Calculated creatinine clearance

  * ≥ 30 cc/min using the Cockcroft-Gault formula (Cockcroft and Gault 1976)
  * or by equivalent criteria such as measured GFR by hospital's laboratory
  * or by 24-hour urine collection for determination of creatinine clearance:

Males:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) . 72 x serum creatinine (mg/dL)

Females:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)

Hepatic:

* Bilirubin ≤ 1.5 × upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 × ULN
* Alanine aminotransferase (ALT) ≤ 2.5 × ULN

Coagulation:

* International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤ 1.5× ULN for patients who are not on any anticoagulants.

Patients who are on warfarin would require switching to either a short acting anticoagulant such as oral apixaban or lovenox injection. Prior to entry on the trial their INR should be <2.0. Patients who are already on short acting anticoagulants would be allowed to enroll on the study provided their INR <2.0

* Females of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to registration.
* Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use a highly effective method of contraception from the time of informed consent until 90 days after treatment discontinuation.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.
* Availability of baseline tumor tissue (fresh biopsy or archival) prior to enrollment on the clinical trial. TURBT specimens are preferred but tissue from lymph node or visceral areas are also acceptable. If archival tissue is not available, the subject must be willing to consent to a fresh biopsy for research prior to registration for protocol therapy. If archival tissue is not available and there are no sites amenable to biopsy, enrollment must be discussed with the sponsor-investigator on a case by case basis.
* Palliative radiation therapy prior to or during the treatment is allowed if indicated. However, if prior to start of treatment, radiation therapy must complete at least 7 days prior to cycle 1 day 1 of treatment.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Participation in another clinical study with an investigational product within 2 weeks prior to registration.
* Any previous treatment with a PD1 or PD-L1 inhibitor, including Avelumab.
* Previous systemic immunotherapy. Previous use of intravesical BCG is acceptable.
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence. However adequately treated prostate cancer >3 years ago with no significant change in PSA for past 6 months can be included.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ.
* Receipt of the last dose of anti-cancer therapy for local recurrence only and not for any systemic disease (immunotherapy, endocrine therapy, biologic therapy, tumor embolization, monoclonal antibodies, or other investigational agent) within14 days prior to study registration and within 6 weeks for intravesical BCG or mitomycin C .
* Mean QT interval corrected for heart rate (QTc) ≥470 ms on electrocardiogram (ECG) using Frediricia's Correction.
* Current or prior use of immunosuppressive medication within 28 days before study registration, with the exceptions of: a) intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection) b) systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid, c) steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Any unresolved toxicity (≥CTCAE grade 2) from previous anti-cancer therapy. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss). Alopecia, sensory neuropathy grade ≤ 2, or other grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
* Active or prior documented autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. NOTE: Subjects with diabetes type I, vitiligo, hypo- or hyperthyroid diseases, or psoriasis not requiring immunosuppressive systemic treatment are eligible. Patients with a history of completely resolved childhood asthma or atopy are also eligible.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of and/or confirmed pneumonitis.
* History of primary immunodeficiency.
* History of organ transplantation including allogeneic stem-cell transplant.
* History of hypersensitivity to Avelumab or Eribulin mesylate, including known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3).
* Uncontrolled intercurrent illness including, but not limited to:

  * ongoing or active infection requiring systemic therapy
  * active peptic ulcer disease or gastritis, or active bleeding diatheses,
  * psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Any subject known to have evidence of acute or chronic hepatitis B (positive HBV surface antigen), hepatitis C (perform HCV RNA if anti-HCV antibody screening test positive), or human immunodeficiency virus (HIV). Note: testing will be performed if applicable per physician discretion.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of starting treatment with Avelumab. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control. For this study male or female patients of reproductive potential need to employ two highly effective and acceptable forms of contraception throughout their participation in the study and for 90 days after last dose of study drug.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Brain metastases or history of leptomeningeal carcinomatosis.
* Subjects with uncontrolled seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monika Joshi, M.D., Study Chair — Big Ten Cancer Research Consortium
Locations (2):
- United States (2):
  - Univeristy of Iowa Hospital and Clinics, Iowa City, Iowa
  - Penn State Cancer Intsitute, Hershey, Pennsylvania

REFERENCES:
- [Derived] Joshi M, Holder SL, Zhu J, Zheng H, Komanduri S, Warrick J, Yasin H, Garje R, Jia B, Drabick JJ, DeGraff DJ, Zakharia Y. Avelumab in Combination with Eribulin Mesylate in Metastatic Urothelial Carcinoma: BTCRC GU-051, a Phase 1b Study. Eur Urol Focus. 2022 Mar;8(2):483-490. doi: 10.1016/j.euf.2021.03.005. Epub 2021 Mar 17. PMID 33741296
- See also: Big Ten Cancer Research Consortium Website — http://www.bigtencrc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 0: Starting Cohort: Eribulin mesylate: 1.1mg/m2 on days 1,15 Avelumab 10 mg/kg on days 1,15
- Dose Level 1: Eribulin mesylate 1.4mg/m2 days 1,15 Avelumab 10mg/kb on days 1,15
Period: Overall Study
Arm/Group | Dose Level 0: Starting Cohort | Dose Level 1
Started | 3 | 3
Completed | 0 | 1
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Disease Progression | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 0: Starting Cohort | Dose Level 1 | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (8.5) | 69.3 (9.1) | 70.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
Smoking Status [Count of Participants; unit: Participants]
  Never a smoker | 3 | 1 | 4
  Former smoker | 0 | 2 | 2
Histology [Count of Participants; unit: Participants]
  Urothelial(transitional cell) Carcinoma | 2 | 2 | 4
  Urothelial(transitional cell) Carcinoma, Mixed | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Assess the Adverse Events of Combining Eribulin Mesylate With Avelumab - (MTD Cohort)
Description: Dose limiting toxicities (DLTs) experienced by subjects while being treated with the combination of eribulin+avelumab, by dose level.
Time Frame: 4-weeks
Measure: Number; unit: participants
Arm/Group | Dose Level 0: Starting Cohort | Dose Level 1
Number analyzed (Participants) | 3 | 3
participants
  Neutrophil Count Decreased | 0 | 1
  Febrile Neutropenia | 0 | 1

2. Primary Outcome: Assess Response Rates (RR) - (Efficacy Cohort)
Description: Complete Response (CR) + Partial Response (PR)
Time Frame: 12 months
Population: Data for this outcome measure was not collected or analyzed due to the early termination of the study.
Arm/Group | Dose Level 0: Starting Cohort | Dose Level 1
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Assess Disease Control Rate (DCR)
Description: Complete Response (CR) + Partial Response (PR) + Stable Disease (SD)
Time Frame: at 3, 6 months
Population: Data for this outcome measure was not collected or analyzed due to the early termination of the study.
Arm/Group | Dose Level 0: Starting Cohort | Dose Level 1
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Estimate Progression Free Survival (PFS)
Description: probability that a patient remains free of progression of disease by modified RECIST 1.1
Time Frame: 12 months
Population: Data for this outcome measure was not collected or analyzed due to the early termination of the study.
Arm/Group | Dose Level 0: Starting Cohort | Dose Level 1
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Estimate Overall Survival (OS)
Description: time from start of treatment, Day 1, to the date of death due to any cause
Time Frame: 12 months
Population: Data for this outcome measure was not collected or analyzed due to the early termination of the study.
Arm/Group | Dose Level 0: Starting Cohort | Dose Level 1
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Estimate Median Progression Free Survival (PFS)
Description: measurement from the date of initiation of avelumab+ eribulin, D1 until the criteria for disease progression is met as defined by modified RECIST 1.1
Time Frame: 12 months
Population: Data for this outcome measure was not collected or analyzed due to the early termination of the study.
Arm/Group | Dose Level 0: Starting Cohort | Dose Level 1
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Estimate Median Overall Survival (OS)
Description: time from start of treatment, Day 1, that half of the patients in the group with the disease are still alive.
Time Frame: 2.5 years
Population: Data for this outcome measure was not collected or analyzed due to the early termination of the study.
Arm/Group | Dose Level 0: Starting Cohort | Dose Level 1
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Assess the Duration of Response
Description: the period measured from the time that measurement criteria are met for complete or partial response (whichever status is recorded first) until the date that recurrent or progressive disease is objectively documented.
Time Frame: 2.5 years
Population: Data for this outcome measure was not collected or analyzed due to the early termination of the study.
Arm/Group | Dose Level 0: Starting Cohort | Dose Level 1
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to six cycles (6 months)
Groups:
- All Subjects: All subjects (6) from each dose level.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=6)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
FEVER (General disorders) | 1 (1)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=6)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 3 (6)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CHILLS (General disorders) | 3 (3)
CREATININE INCREASED (Investigations) | 3 (3)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1)
EDEMA LIMBS (General disorders) | 1 (2)
FATIGUE (General disorders) | 2 (2)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (3)
HYPOTHYROIDISM (Endocrine disorders) | 1 (2)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 1 (2)
INFUSION RELATED REACTION (General disorders) | 2 (2)
INFUSION SITE EXTRAVASATION (General disorders) | 1 (2)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 1 (1)
LIPASE INCREASED (Investigations) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 3 (5)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
NAIL INFECTION (Infections and infestations) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (8)
PARESTHESIA (Nervous system disorders) | 1 (1)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1)
SERUM AMYLASE INCREASED (Investigations) | 1 (2)
SINUS PAIN (Nervous system disorders) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 1 (1)
SURGICAL AND MEDICAL PROCEDURES (Surgical and medical procedures) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (2)
VOMITING (Gastrointestinal disorders) | 2 (2)
WHITE BLOOD CELL DECREASED (Investigations) | 2 (8)

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, no primary or secondary endpoints were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT03502681/Prot_SAP_000.pdf